CLINICAL TRIAL: NCT01818830
Title: Amino Acids Expression Profiling of Patients With Sepsis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Longxiang Su, Attending Doctor, Chinese PLA General Hospital
Other Study IDs: PLAGHHN2013001
Record Dates: First submitted 2013-03-23; First posted 2013-03-27 (Estimated); Last update posted 2013-03-27 (Estimated); Status verified 2013-03

CONDITIONS: Sepsis; Amino Acids
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- SIRS group: (1) temperature > 38oC or < 36oC; (2) pulse rate > 90 beats/min; (3) ventilation rate > 20 breaths/min or hyperventilation with a partial pressure of arterial carbon dioxide (PaCO2) < 32 mmHg; (4) white blood cell (WBC) count >1 2,000μL-1 or < 4000 μL-1 , or > 10% immature cells.
- sepsis: SIRS+infection
- normal control: For the healthy control outpatients, possibilities of acute or past chronic diseases were excluded. Moreover, we made sure that the healthy control subjects had not been hospitalized or taken vitamin-based substitutive drugs in the last 12 months, and proved normal in physical checkups and lab examinations.

SUMMARY:
The patients with sepsis are in the state of hypermetabolism, increased resting energy expenditure, protein and fat catabolism disorder, negative nitrogen balance, insulin resistance, hyperglycemia, and amino acid metabolism disorders. However, it is remain unclear the changes of amino acids expression profiling in sepsis patients. In this study, the investigators has planned to enroll 100 subjects, including 20 cases with systemic inflammatory response syndrome (SIRS), 20 cases with sepsis, 20 cases with severe sepsis and 20 with septic shock. In addition, this study also include 20 normal cases as control. The serum sample of patients with sepsis is draw on days 1, 3, 5, 7, 10, and 14 after first ICU admission. High-performance liquid chromatography and tandem mass spectrometry was used to detect the quantification of amino acids. The amino acids expression profiling contain Arginine, Ornithine, Histidine, Cystine, Isoleucine, Cystathionine, Leucine, Homocystine, Lysine, α-Amino-n-Butyric Acid, Methionine, Alanine, Phenylalanine, Anserine, Threonine, β-Alanine, Tryptophan, β-Amino-Isobutyric Acid, Valine, Carnosine, γ-Amino-n-Butyric Acid, Ethanolamine, Glycine, δ-Hydroxylysine, Serine, Hydroxy-L-Proline, Taurine, 1-Methyl-L-Histidine, Tyrosine, 3-Methyl-L-Mistidine, α-Amino-Adipic, Phospho-Ethanolamine, Asparagine, Phospho-L-Serine, Aspartic acid, Proline, Citrulline, Sarcosine, Glutamic acid, Argininosuccinic Acid, Glutamine, Homocitrulline. The investigators speculate that measurement of amino acids expression profiling could be taken as an indicator for assessment in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female aged 18 years old and over;
2. Clinically confirmed infection;
3. Fulfilled at least two criteria of systemic inflammatory response syndrome (a) core temperature higher than 38 °C or lower than 36 °C (b)respiratory rate above 20/min, or PCO2 below 32 mmHg (c) pulse rate above 90/min, and (d) white blood cell count greater than 12,000/μl or lower than < 4,000/μl or less than 10% of bands.

Exclusion Criteria:

1. parenteral nutrition;
2. diabetes and other metabolic-related diseases;
3. chronic liver disease;
4. neutropenia (≤ 500 neutrophils/mm3);
5. HIV infection;
6. patients or their relatives refused.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The inpatients were included who were in the intensive care units (ICU) of the Department of Respiratory Disease, the Emergency Department, and the Department of Surgery of the Chinese People's Liberation Army General Hospital from March 2012.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Patients Outcome | 28 days
  The survival time of patients more than 28 days is defined as survival. The survival time of patients less than 28 days is defined as death.

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Xie, Doctor, Study Director — Department of Respiratory Diseases, Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Su L, Li H, Xie A, Liu D, Rao W, Lan L, Li X, Li F, Xiao K, Wang H, Yan P, Li X, Xie L. Dynamic changes in amino acid concentration profiles in patients with sepsis. PLoS One. 2015 Apr 7;10(4):e0121933. doi: 10.1371/journal.pone.0121933. eCollection 2015. PMID 25849571